CLINICAL TRIAL: NCT04039061
Title: Autosomal Dominant Polycystic Kidney Disease Patient Registry
Brief Title: ADPKD Patient Registry
Acronym: ADPKD
Status: Recruiting | Type: Observational
Sponsor: PKD Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 120190065
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADPKD patients: Patients with a diagnosis, or suspected diagnosis, of ADPKD

SUMMARY:
The purpose of the ADPKD Registry is to create an online patient network that includes at least 5,000 people with Autosomal Dominant Polycystic Kidney Disease (ADPKD) who contribute data on their health and other topics. The ADPKD Patient Registry aims to support important scientific discoveries and support patient needs in the following ways:

* Connect ADPKD patients with opportunities to join clinical studies.
* Collect data for the research community to better describe the ADPKD disease experience and improve patient care.
* Engage with patients by measuring quality of life outcomes.

DETAILED DESCRIPTION:
The ADPKD Registry will be a patient-powered network of people with ADPKD. This data will inform new research to improve ADPKD patient outcomes, learn more about the patient journey and discover unmet medical needs. We collect data most relevant to your ADPKD diagnosis, its major symptoms and management, as well as key demographic data (no personally identifiable information is shared). A Registry keeps information in one place making it easier for researchers to utilize Registry information while still protecting the privacy of those who take part. The Registry will be hosted on a secure, online platform that patients can access using their home computers, tablets or phones.

The purpose of the ADPKD Registry is to allow PKD patients to:

* Connect with researchers and express interest in taking part in certain clinical studies for ADPKD, including studies of new medications and other treatments.
* Take confidential health-related surveys. These surveys are aimed at better understanding of the health of people with PKD across their lifespans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or suspected diagnosis with autosomal dominant polycystic kidney disease (ADPKD)

Exclusion Criteria:

* caretakers, family members or friends of individuals with ADPKD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone with ADPKD, or suspects that they have ADPKD, is welcome to participate
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2029-09-04 (Estimated); Study Completion 2029-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of people with polycystic kidney disease who experience health-related quality-of-life changes | 1 year
  To be assessed with online modules, developed both internally and through validated partners

CONTACTS AND LOCATIONS:
Overall Officials: Chris Rusconi, PhD, Principal Investigator — PKD Foundation
Locations (1):
- PKD Foundation, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided